CLINICAL TRIAL: NCT03745599
Title: Evaluation of the Effects of Different Analgesics on Pain and Health-related Quality of Life of Patients With Pericoronitis in the Short-term Period: A Randomized, Double-blind, Clinical Trial
Brief Title: Evaluation of the Effects of Different Analgesics on Pericoronitis Pain and Quality of Life
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, abdullah alalwani, Research Assistant, Near East University, Turkey
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Near East Uni
Record Dates: First submitted 2018-11-13; First posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Pain; Quality of Life
Keywords: Pericoronitis; Analgesics; Non steroid anti-inflammatory drugs; Benzydamine; Quality of life
MeSH Terms: conditions — Pain; Pericoronitis | interventions — Diclofenac; Flurbiprofen; Benzydamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diclofenac (Experimental): Diclofenac group, which received diclofenac 50 mg capsules (Cataflam) and placebo sprays. Placebo sprays have consisted of a normal saline solution and peppermint flavor.
  Interventions: Drug: Diclofenac
- Flurbiprofen (Experimental): Flurbiprofen group, which received flurbiprofen 100 mg capsules and placebo sprays. Placebo sprays have consisted of a normal saline solution and peppermint flavor.
  Interventions: Drug: Flurbiprofen
- Benzydamine (Experimental): Benzydamine group, which received benzydamine 0.045 g, 30 mL oral sprays (Tantum Verde) and placebo capsules. Placebo capsules contained starch.
  Interventions: Drug: Benzydamine

INTERVENTIONS:
Drug: Diclofenac — All patients were instructed to take one capsule orally every 8 h and apply the spray (4 puffs to the pericoronitis area) every 4 h for 7 days, commencing immediately after the clinical examination.
  Arms: Diclofenac
Drug: Flurbiprofen — All patients were instructed to take one capsule orally every 8 h and apply the spray (4 puffs to the pericoronitis area) every 4 h for 7 days, commencing immediately after the clinical examination.
  Arms: Flurbiprofen
Drug: Benzydamine — All patients were instructed to take one capsule orally every 8 h and apply the spray (4 puffs to the pericoronitis area) every 4 h for 7 days, commencing immediately after the clinical examination.
  Arms: Benzydamine

SUMMARY:
Pericoronitis is a painful inflammatory condition which is well known for its negative impact on quality of life of those affected. The aim of this study was to test two hypotheses: (1) that topical application of Benzydamine is as effective as oral Diclofenac or Flurbiprofen in improving pain and quality of life of patients with pericoronitis and (2) that there would be no difference between the effects of the two oral NSAIDs on pain and quality of life of patients with pericoronitis

ELIGIBILITY:
Inclusion Criteria:

* Young adults aged 18 years or over
* Diagnosed with mild pericoronitis
* Having semi-impacted mandibular third molar
* Symptoms of pain and localized swelling

Exclusion Criteria:

* Smoking
* History of allergy to diclofenac, flurbiprofen, benzydamine or other NSAIDs
* Use of systemic antibiotics or analgesics within 3 days before admission
* The patients who had symptoms of severe pericoronitis such as fever higher than 101°F, dysphagia, trismus or facial swelling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-09-03 (Actual); Study Completion 2018-11-02 (Actual)

PRIMARY OUTCOMES:
Oral Health-Related Quality of Life Scores Evaluated | Baseline
  For the pre- treatment period, the Oral Health-Related Quality of Life scores change was evaluated in the 1st day after the clinical examination and before the treatment with the help of the 5-point Likert-type scale where each item was scored from 1 (no trouble) to 5 (lots of trouble).
Oral Health-Related Quality of Life Scores Evaluated | one week after drug prescribed
  For the post - treatment period, the Oral Health-Related Quality of Life scores change was evaluated with the help of the 5-point Likert-type scale where each item was scored from 1 (no trouble) to 5 (lots of trouble). Evaluated periods were 1, 2, 3, 5 and 7 days

SECONDARY OUTCOMES:
Pain Scores Evaluated | Baseline
  For the pre-treatment period, the pain scores change was evaluated in the 1st day after the clinical examination and before the treatment with the help of the visual analog scale (VAS) ranging from 0 (no pain) to 10 (most severe pain).
Pain Scores Evaluated | one week after drug prescribed
  For the post-treatment period, the pain scores change was evaluated in the 1, 2, 3, 5 and 7days with the help of the visual analog scale (VAS) ranging from 0 (no pain) to 10 (most severe pain).

OTHER OUTCOMES:
Oral Health Impact Profile (OHIP-14) Scores Evaluated | Baseline and one week after drug prescribed
  Before and after the treatment period, the Oral Health Impact Profile scores change was evaluated in the 1st day after the clinical examination and before the treatment (baseline), and after 7 days with the help of the 5-point scale where each item was scored from "never" = 0, "hardly ever" = 1, "occasionally" = 2, "fairly often" = 3, "very often = 4"

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah AlAlwani, DDS, Principal Investigator — Near East University
Locations (1):
- Abdullah AlAlwani, Mersin, Turkey (Türkiye)